CLINICAL TRIAL: NCT05029869
Title: Monitoring Minimal Residual Disease in Gastric Cancer by Liquid Biopsy
Brief Title: Monitoring Minimal Residual Disease in Gastric Cancer by Liquid Biopsy Study Description
Status: Active, not recruiting | Type: Observational
Sponsor: University Medical Center Ho Chi Minh City (UMC) (Other)
Responsible Party: Sponsor
Other Study IDs: 81/GCN-HDDD 2021
Record Dates: First submitted 2021-08-25; First posted 2021-09-01 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-06

CONDITIONS: Gastric Cancer; ctDNA
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: ctDNA — The blood samples for ctDNA and other tumor markers will be first collected within 14 days before surgery, and then be tested after gastrectomy in scheduled interval

SUMMARY:
This study aims to evaluate the use of Next Generation Sequencing (NGS) to detect circulating tumor DNA in gastric cancer patients after gastrectomy

DETAILED DESCRIPTION:
Gastric cancer is the fourth most common cancer in Vietnam with high mortality rate. Patients at early stages undergo radical gastrectomy with curative intent, but the remaining tumor cells, termed as minimal residual disease (MRD), can later cause relapse. Conventional methods to monitor MRD such as imaging and blood tests for biomarkers such as CEA are not sensitive and specific enough. ctDNA has recently emerged as a promising noninvasive marker with high accuracy to monitor MRD and detect relapse in many cancers such as breast and colorectal cancers. However, its application in gastric cancer has not been extensively evaluated. Therefore, this study aims to use advanced NGS technologies to detect ctDNA in liquid biopsy as a biomarker to monitor MRD after radical gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female patients aged 18 years and older
2. Histologically proven primary gastric adenocarcinoma before surgery
3. Clinical stage is locally advanced cT2-4a any N and M0
4. In initial evaluation, patient can undergo radical gastrectomy and lymphadenectomy
5. No preoperative therapy, including chemotherapy and radiotherapy
6. No known cancer diagnosis within last five years
7. Signed informed consent

Exclusion Criteria:

1. Gastrectomy cannot be achieved during operation due to metastasis
2. Patient fails to follow-up and provide postoperative samples

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed and untreated gastric adenocarcinoma
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-10-04 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
The sensitivity of MRD detection using ctDNA as the biomarker | 2 years after surgery
  The percentage of positive ctDNA detection among participants who experience disease recurrence or metastasis
The specificity of MRD detection using ctDNA as the biomarker | 2 years after surgery
  The percentage of positive ctDNA detection among participants who do not experience disease recurrence or metastasis

SECONDARY OUTCOMES:
Leading time between ctDNA detection and cancer recurrence detected by conventional methods | 2 years after surgery
  Time is measured between first positive ctDNA detection and first cancer recurrence detected by conventional methods
Mean ctDNA level (MTM/ml) of gastric cancer before operation | Within 14 days before operation
  The mean ctDNA level in gastric cancer patients before operation
Mutation profile of gastric cancer | Within 14 days before operation
  Profiling of the most frequent gene mutations

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Ho Chi Minh City, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No